CLINICAL TRIAL: NCT05093647
Title: Sexual Function Changes in High-Risk Pregnancies
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sevim Özge Özdemir, perinatology specialist, Saglik Bilimleri Universitesi
Other Study IDs: FSFI
Record Dates: First submitted 2021-10-03; First posted 2021-10-26 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Sexual Dysfunctions, Psychological; High Risk Pregnancy; Sexual Behavior
Keywords: sexual dysfunction, high-risk pregnancy, FSFI, quality of life
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Behavior; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient: The women who followed up for HrP (high-risk pregnancy ) were invited to participate and women with HrP in the second trimester (14th to 28th gestational weeks), between 20 to 40 years old, and followed up at our perinatology department with a diagnosis of IUGR (intrauterine growth retardation
  ), cholestasis, diabetes, preeclampsia, or hypertension were included.
- control: The pregnant women admitted for routine second-trimester ultrasonography assessment but with no risk for pregnancy formed the control group.

SUMMARY:
Sexual Function Changes in High-Risk Pregnancies

DETAILED DESCRIPTION:
Background and Aim: Sexual functions generally decrease during pregnancy, and high-risk pregnancies are more severe clinical conditions that cause couples to reduce or abstain entirely from their intimacy. However, the evidence on the sexual functions in high-risk pregnancies is scarce. Therefore, this study aimed to evaluate the sexual function changes in high-risk pregnancies compared to normal pregnancies.

Methods: A total of 200 pregnant women (100 women in high-risk pregnancy and normal pregnancy groups each) were included. Demographic and obstetric data were collected, and participants completed The Female Sexual Function Index (FSFI).

ELIGIBILITY:
Inclusion Criteria:

study grup Pregnant women who ; followed up for HrP in the second trimester (14th to 28th gestational weeks), between 20 to 40 years old, followed up at our perinatology department with a diagnosis of IUGR, cholestasis, diabetes, preeclampsia, fetal anomaly control grup admitted for routine second-trimester ultrasonography assessment but with no risk for pregnancy

Exclusion Criteria:

Pregnant women who ; younger than 20 or older than 40 years of age, gestation in the 1st or 3rd trimester, presence of psychiatric or chronic disorders like rheumatic or heart diseases,

-

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The women who followed up for HrP were invited to participate and women with HrP in the second trimester (14th to 28th gestational weeks), between 20 to 40 years old, and followed up at our perinatology department with a diagnosis of IUGR, cholestasis, diabetes, preeclampsia, or hypertension were included.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Sexual dysfunction rate in high risk pregnancies | 3 month
  Sexual dysfunction rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Maternal-Fetal Medicine Unit, Başakşehir City Hospital, Hamidiye School of Medicine, University of Health Sciences,, Başaksehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McCool ME, Zuelke A, Theurich MA, Knuettel H, Ricci C, Apfelbacher C. Prevalence of Female Sexual Dysfunction Among Premenopausal Women: A Systematic Review and Meta-Analysis of Observational Studies. Sex Med Rev. 2016 Jul;4(3):197-212. doi: 10.1016/j.sxmr.2016.03.002. Epub 2016 Apr 19. PMID 27871953
- [Result] Alizadeh S, Riazi H, Alavi-Majd H, Ozgoli G. Prevalence of female sexual dysfunction during pregnancy in Eastern Mediterranean Regional Office Countries (EMRO): a systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2022 Dec;35(25):6654-6662. doi: 10.1080/14767058.2021.1919074. Epub 2021 May 4. PMID 33944668
- [Result] Sartorao Filho CI, Pinheiro FA, Prudencio CB, Nunes SK, Takano L, Enriquez EMA, Orlandi MIG, Junginger B, Hallur RLS, Rudge MVC, Barbosa AMP. Impact of gestational diabetes on pelvic floor: A prospective cohort study with three-dimensional ultrasound during two-time points in pregnancy. Neurourol Urodyn. 2020 Nov;39(8):2329-2337. doi: 10.1002/nau.24491. Epub 2020 Aug 28. PMID 32857893